CLINICAL TRIAL: NCT07257510
Title: A Prospective, Multicenter Clinical Study of Pomalidomide Combined With Orelabrutinib and Zuberitamab in Treatment-Naive Mantle Cell Lymphoma
Brief Title: Pomalidomide Plus Orelabrutinib and Zuberitamab in Untreated Mantle Cell Lymphoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POZ
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-08

CONDITIONS: Mantle Cell Lymphoma (MCL); POZ
MeSH Terms: conditions — Lymphoma, Mantle-Cell | interventions — pomalidomide; orelabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pomalidomide + Orelabrutinib + Zuberitamab and Orelabrutinib + Zuberitamab Maintenance (Experimental): 1. In induction phase, patients will receive pomalidomide 4mg/day PO once daily day1-12/cycle; orelabrutinib 150 mg/day PO once daily; and zuberitamab 375 mg/m² IV on day 1/cycle, every 28 day per cycle for 6 cycles. 2. In maintenance phase, Patients with MRD negative (≤10-5) after induction therapy will recieve orelabrutinib 150 mg/day PO once daily for 18cycles and zuberitamab 375 mg/m² IV on day 1 of cycle 7, 10, 13, 16, 19 and 22, every 28 day per cycle.
  Interventions: Drug: Pomalidomide; Drug: Orelabrutinib; Drug: Zuberitamab

INTERVENTIONS:
Drug: Pomalidomide — 4mg/day PO once daily, day1-21/cycle
  Other Names: Induction phase
Drug: Orelabrutinib — 150mg/day PO once daily
  Other Names: Induction phase
Drug: Zuberitamab — 375 mg/m² IV on day 1/cycle
  Other Names: Induction phase
Drug: Zuberitamab — 375 mg/m² IV on day 1 of cycle 7, 10, 13, 16, 19 and 22,
  Other Names: Maintenance phase

SUMMARY:
This multicenter trial evaluates the efficacy and safety of pomalidomide combined with orelabrutinib and zuberitamab (POZ) in patients with mantle cell lymphoma (MCL). After six cycles of POZ, patients who achieved minimal residual disease (MRD) negativity received maintenance therapy with orelabrutinib plus zuberitamab for up to 18 cycles. Those with MRD positivity were excluded and received alternative treatments. The primary endpoint is the MRD rate after six cycles of POZ. Secondary endpoints include progression-free survival (PFS), overall survival (OS), MRD rate, objective response rate (ORR), and safety.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed mantle cell lymphoma
* Age 18-80 years, both genders are eligible..
* Untreated MCL.
* At least one measurable lesion. Measurable disease is defined as a tumor mass measurable in one or two dimensions ≥1.5 cm, as well as measurable spleen lesions.
* Any one of the following factors is present:: MIPI intermediate-high risk, ki67≥30%, blastoid/pleomorphic, TP53 abnormality (mutation/deletion) or p53 protein expression >50%, large mass (maximum diameter ≥7.5cm), complex karyotype (≥3 chromosomal abnormalities (excluding t(11; 14)))
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 2.
* Hematologic function is adequate, defined as:

  1. Absolute neutrophil count (ANC) ≥1×109/L, growth factor support must not be used within 7 days prior to testing;
  2. Platelet count ≥75×10⁹/L, or ≥50×10⁹/L (if bone marrow involvement), no use of growth factor support or transfusion allowed within 7 days prior to testing.
* Adequate hepatic function per local laboratory reference range as follow:

  1. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5× the upper limit of normal (ULN);
  2. Bilirubin ≤ 2 × ULN (except for those diagnosed with Gilbert's syndrome, which allows up to 5 × ULN)
* Adequate renal function as demonstrated by:

  1. Creatinine clearance ≥60 mL/min (estimated using the Cockcroft-Gault formula or the glomerular filtration rate [eGFR] estimated using the Modification of Diet in Renal Disease [MDRD] formula)
  2. Serum creatinine ≤1.5×ULN
* International Normalized Ratio (INR) ≤ 1.5 × ULN and Activated Partial Thromboplastin Time (APTT) ≤ 1.5 × ULN
* Life expectancy of more than 3 months.
* Ability to provide written informed consent and understand and comply with study requirements.
* Able to comply with the study visit schedule and other protocol requirements

Exclusion Criteria:

* Current central nervous system involvement or suspected patients and those with a history of this condition
* Previously received systemic treatment for MCL, including BTKi.
* Uncontrolled active systemic fungal, bacterial, or viral infections (defined as persistent signs/symptoms related to the infection despite the use of appropriate antibiotics, antiviral therapy, and/or other treatments with no improvement).
* Known human immunodeficiency virus (HIV) infection, or the following serological status indicating active hepatitis B or C virus infection:

  1. Subjects with positive hepatitis B virus core antibody (HBcAb) and negative surface antigen (HBsAg) must have a negative polymerase chain reaction (PCR) result prior to the first dose. Subjects with positive HBsAg or HBV-DNA:
  2. Subjects with positive hepatitis C antibodies must have an HCV-RNA negative result before the first dose. Subjects with positive hepatitis C PCR results will not be eligible for this study.
* Clinically severe cardiovascular diseases, including:

  1. Myocardial infarction occurring within the 6 months prior to screening;
  2. Unstable angina occurring within 3 months prior to screening;
  3. Clinically significant arrhythmias (e.g., sustained ventricular tachycardia, ventricular fibrillation, torsades de pointes ventricular tachycardia);
  4. QTcF (corrected by Fridericia's formula) > 480 msec;
  5. History of second-degree type II atrioventricular (AV) conduction block or third-degree atrioventricular conduction block;
  6. III or IV congestive heart failure as defined by the New York Heart Association (NYHA)
* History of severe hemorrhagic disorders, such as hemophilia A, hemophilia B, von Willebrand disease, or a history of spontaneous bleeding requiring blood transfusion or other medical interventions.
* History of deep vein thrombosis (DVT) or pulmonary embolism (PE) in the past 12 months
* History of significant cerebrovascular disease/events within 6 months prior to the first administration of the investigational drug, including stroke or intracranial hemorrhage.
* Unable to swallow capsules or having significant gastrointestinal functional disorders, such as malabsorption syndrome, gastric or small intestine resection, symptomatic inflammatory bowel disease, or partial or complete intestinal obstruction.
* Continuous treatment with strong and moderate CYP3A inhibitors or CYP3A inducers is required. If the patient has taken strong or moderate CYP3A inhibitors or inducers within 7 days prior to the first dose of the investigational drug (or has taken these drugs for less than 5 half-lives), they cannot be enrolled. Patients using moderate CYP3A inhibitors can be considered for the study after at least a 7-day washout period.
* Anticoagulation treatment with warfarin or equivalent vitamin K antagonists (e.g., phenprocoumon) is required within 7 days after the first dose of the investigational drug or receiving anticoagulation therapy.
* Pregnant or breastfeeding women
* Hypersensitivity to any investigational drug
* Any mental or cognitive impairment that may limit their understanding, execution, and compliance with the informed consent form and the study.
* Subjects with drug abuse and alcoholism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Minimum residual disease (MRD) rate | 6 months
  After 6 cycles of the pomalidomide combined with orelabrutinib and zuberitamab (POZ) regimen, the proportion of patients with undetectable minimal residual disease (MRD) (≤10-5) as evaluated by the high-throughput sequencing (NGS) platform.

SECONDARY OUTCOMES:
MRD rate | 3 months
  The proportion of patients with undetectable minimal residual disease (MRD) (≤10-5) as evaluated by the high-throughput sequencing (NGS) platform.
MRD rate | 12 months
  The proportion of patients with undetectable minimal residual disease (MRD) (≤10-5) as evaluated by the high-throughput sequencing (NGS) platform.
MRD rate | 18 months
  The proportion of patients with undetectable minimal residual disease (MRD) (≤10-5) as evaluated by the high-throughput sequencing (NGS) platform.
MRD rate | 24 months
  The proportion of patients with undetectable minimal residual disease (MRD) (≤10-5) as evaluated by the high-throughput sequencing (NGS) platform.
Overall Response Rate | up to 3 years
  Percentage of participants with overall response was determined on the basis of investigator assessments according to 2014 Lugano criteria.
Progression-free survival | up to 3 years
  Progression-free survival was defined as the time from the date of randomization until the date of the first documented day of disease progression or relapse, using 2014 Lugano criteria, or death from any cause, whichever occurred first.
Overall survival | up to 3 years
  Overall survival was defined as the time from the date of randomization to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No